CLINICAL TRIAL: NCT01411358
Title: Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine, Formulation 2011-2012, in Non-Elderly Adult and Elderly Subjects
Brief Title: Immunogenicity and Safety of AdimFlu-S 2011-2012 in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLU11T12A
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: influenza; vaccine; immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdimFlu-S 2011-2012 (Experimental)
  Interventions: Biological: non-elderly aged between 18 and 60; Biological: elderly aged over 60

INTERVENTIONS:
Biological: non-elderly aged between 18 and 60 — one dose of 0.5mL AdimFlu-S
Biological: elderly aged over 60 — one dose of 0.5mL AdimFlu-S

SUMMARY:
The purpose of this study is to evaluate the antibody response to each of the three influenza vaccine strains included in the licensed seasonal flu vaccine, as measured by hemagglutination inhibition (HAI) at 21 days post immunization in non-elderly and elderly subjects in compliance with the requirements of the current European Union (EU) recommendations for the evaluation of the immunogenicity for a new formulation of a licensed flu vaccine (CPMP/BWP/214/96).

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females and aged ≥ 18 years;
* Willing and able to adhere to visit schedules and all study requirements;
* Subjects read and signed the study-specific informed consent.

Exclusion Criteria:

* Subject or his/her family is employed by the participated hospital;
* Subjects received 2010-2011 seasonal influenza vaccine within the previous 6 months;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication
* Personal or family history of Guillain-Barré Syndrome
* An acute febrile illness within 1 week prior to vaccination;
* Current upper respiratory illness, including the common cold or nasal congestion within 72 hours
* Subjects with influenza-like illness as defined by the presence of fever (temperature ≥ 38°C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough
* Female subjects who are pregnant during the study
* Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent
* Immunodeficiency, or under immunosuppressive treatment
* Receipt of any vaccine within 1 week prior to study vaccination or expected receipt between Visit 1 (study vaccination) and Visit 2 (final collection of blood samples);
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the seroprotection rate which is defined as the proportion of subjects with HAI titer ≥ 40. | 3 weeks post vaccination
  Serum samples will be tested for anti-hemagglutinin (HA) antibodies by hemagglutination inhibition (HAI).

CONTACTS AND LOCATIONS:
Overall Officials: Gin-Hsiang Wu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan